CLINICAL TRIAL: NCT01989507
Title: Very Low-Nicotine Cigarettes in Smokers With SUD: Smoking, Substance Use Effects
Brief Title: Very Low-Nicotine Cigarettes in Smokers With SUD
Acronym: VLNC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Damaris J. Rohsenow, Ph.D., Principal Investigator, Brown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01DA034628-01A1 (NIH)
Record Dates: First submitted 2013-11-12; First posted 2013-11-21 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Nicotine Dependence
Keywords: tobacco smoking; smoking cessation; nicotine dependence; tobacco use disorder
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Smoking; Smoking Cessation | interventions — Nicotine; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Very low nicotine content cigarettes (Experimental): Cigarettes with Nicotine Yield 0.07 ± 0.02
  Interventions: Drug: Nicotine; Behavioral: behavioral counseling for smoking cessation
- Conventional nicotine content cigarettes (Active Comparator): Cigarettes with Nicotine Yield 0.8 ± 0.15
  Interventions: Drug: Nicotine; Behavioral: behavioral counseling for smoking cessation

INTERVENTIONS:
Drug: Nicotine
Behavioral: behavioral counseling for smoking cessation — Brief session of Brief advice. Assess smoking and provide assistance with quitting via coping skills.

SUMMARY:
The purpose of this study is to determine the efficacy, acceptability and unintended consequences of very low nicotine content cigarettes (VLNCC) in smokers with current or past year substance use disorders (SUD). The primary aim of this study is to determine whether 6 weeks of VLNCC compared to normal nicotine content cigarettes (NNCC) will result in more smoking cessation over 6 months and reduce cigarette use, cotinine, and biomarkers of toxicity. We will also assess the effects of VLNCC versus NNCC cigarettes on frequency of substance use and substance cravings (drugs and alcohol) because this is relevant to the safety of these products among smokers with SUD. Secondary aims are to study effects on cigarette craving, nicotine withdrawal and dependence, and depressed mood. Methods: Random assignment to VLNCC versus NNCC of up to 312 smokers with SUD will be balanced by gender, degree of tobacco dependence, and recent drug and alcohol use. All smokers will be provided with smoking counseling. Assessments over 6 months will assess effects both during the 6 weeks of using research cigarettes and after return to usual cigarettes. The importance is in determining the viability and safety of this public health strategy in terms of effects on both smoking and other substance use in a highly addicted population, which is essential to determine before the FDA implements this policy.

DETAILED DESCRIPTION:
The 2009 passage of the Family Smoking Prevention and Tobacco Control Act (FSPTCA) gave the Food and Drug Administration (FDA) the authority to reduce levels of nicotine in cigarettes if appropriate for public health. This project addresses an area targeted for study by NIH and the FDA to assess the impact of products with reduced toxicity on tobacco use behaviors. Very-low nicotine content cigarettes (VLNCC) have been shown in some studies with smokers from the general population to reduce craving and withdrawal for tobacco relative to abstinence with little or no compensatory smoking, suggesting that a mandated reduction in the nicotine yield of cigarettes could substantially reduce smoking rates. This may be a particularly effective method of reducing smoking and smoking-related disease in special populations that have very high rates of tobacco dependence, such as people with substance use disorders (SUD). However, the consequences of this policy for smokers with SUD have not been investigated, and a call has gone out for studies of the safety of these products with vulnerable populations such as these. The purpose of this study is to determine the efficacy, acceptability and unintended consequences of VLNCC in smokers with SUD (current or past year) currently abstinent from hard drugs. The primary aims are to determine whether VLNCC will increase smoking cessation and reduce cigarette use, cotinine, and biomarkers of toxicity in smokers with SUD relative to baseline and to those randomized to a normal nicotine content cigarette (NNCC), and to determine any unintended effects of VLNCC on substance use and cravings to use substances so as to investigate safety. Secondary aims are to study effects on cigarette craving and nicotine withdrawal and dependence (mechanisms), and state depression (safety). A 2-group between-group by pre-post design will compare 6 weeks of VLNCC to NNCC; all smokers will also be provided with smoking counseling. Follow-up over 6 months will assess effects after return to usual cigarettes. The importance is in determining the viability and safety of this public health strategy in terms of effects on both smoking and other substance use in a highly addicted population, which is essential to determine before the FDA implements this policy.

ELIGIBILITY:
Inclusion Criteria::

* Diagnostic and Statistical Manual-5 criteria for current or past year substance use disorder
* smoke 10+ cigarettes/day for past 6 months
* zero breath alcohol, negative urine drug tests and a self-report of no drug use in the past 30 days on day of informed consent
* score of 4-8 on the Contemplation Ladder (individuals interested in quitting smoking someday and/or have thought about quitting)

Exclusion Criteria:

* active psychosis as evidenced by hallucinations or delusions
* actively quitting smoking or current use of any nicotine replacement or other smoking cessation treatment
* medication contraindications for smoking cessation (smoking cessation may change the bioavailability of antipsychotics, warfarin, theophylline and insulin)
* other medications that could affect smoking (naltrexone, buprenorphine, acamprosate, anti-seizure medications, disulfiram)
* if on psychotropic medications, not stabilized on psychotropic medications (i.e., anti-depressant, anti-anxiety or anti-manic medications changed within past 4 weeks)
* inability to understand informed consent in a test (true-false questions) on the key elements of the consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
7-day point-prevalence smoking abstinence | 6 weeks
  self-report of past 7 days abstinence confirmed by expired carbon monoxide (CO) reading of 6 ppm or less

SECONDARY OUTCOMES:
Total N'-nitrosonornicotine (NNAL) | 6 weeks
  Urinary N'-nitrosonornicotine and its glucuronide provide a measure of metabolites of the tobacco-specific carcinogen N'-nitrosonornicotine
Number of cigarettes smoked per day | 6 weeks
  Time Line Follow Back for tobacco use will assess self-reported number of cigarettes smoked each day
Number of substance use days | 6 months
  Time Line Follow Back will assess self-reported number of days of drinking or drug use. Any days of either will be counted as a substance use day.
Change in Beck Depression Inventory | Baseline and 6 weeks
  Beck Depression Inventory will be administered at baseline and 6 weeks to detect any change in depression scores from baseline
Total N'-nitrosonornicotine (NNN) | 6 weeks
  Urinary N'-nitrosonornicotine and its glucuronide provide a measure of metabolites of the tobacco-specific carcinogen N'-nitrosonornicotine
3-hydroxypyrene (3-HOP) | 6 weeks
  Urinary 3-hydroxypyrene and its glucuronide and sulfate provides a measure of a metabolite of pyrene, a biomarker for uptake of carcinogenic polycyclic aromatic hydrocarbons
3-hydroxypropylmercapturic acid (3-HPMA) | 6 weeks
  Urinary 3-hydroxypropylmercapturic acid (3-HPMA) provides a measure of a metabolite of the toxicant acrolein
Total urinary cotinine levels | 6 weeks
  cotinine plus cotinine-glucuronide, assessed via urinalysis
duration of longest tobacco abstinence period | 6 weeks
  Time Line Follow Back (TLFB) for tobacco use will be used to record self-reported tobacco abstinence each day. The longest number of contiguous abstinence days will be recorded.
Questionnaire of Smoking Urges, Brief Form | 6 weeks
  Questionnaire of Smoking Urges, Brief Form assesses strong desire/intention to smoke and anticipating negative-affect relief from smoking. The total score from the 10 items will be used.

OTHER OUTCOMES:
Minnesota Nicotine Withdrawal Scale | 6 weeks
  ratings of 7 nicotine withdrawal symptoms will be combined to form a single score for withdrawal
Penn Alcohol Craving Scale | 6 weeks
  Assessment of craving for alcohol over the previous week. Administered weekly for 6 weeks, the mean of the 6 weeks will be used as the outcome variable.
Drug Craving Questionnaire | 6 weeks
  Adapted from Tiffany's Cocaine Craving Questionnaire to assess craving for any drugs over the previous week. Administered weekly for 6 weeks, the mean of the scores over 6 weeks will be used as the outcome variable.
Change in Contemplation Ladder | Baseline and 6 weeks
  The 10-point Contemplation Ladder provides a single continuous measure of motivation to quit smoking. Change from baseline to 6 weeks will be used as the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Damaris J Rohsenow, PhD, Principal Investigator — Brown University; Rosemarie A Martin, PhD, Study Director — Brown University
Locations (1):
- Brown University's Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States